CLINICAL TRIAL: NCT03962712
Title: A Natural Experiment Evaluating the Effect of a Minimum Wage Increase on Obesity and Diet-related Outcomes
Acronym: wages
Status: Completed | Type: Observational
Sponsor: University of Connecticut (Other)
Responsible Party: Principal Investigator, Caitlin Caspi, Associate Professor, University of Connecticut
Other Study IDs: H20-0087
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Nutrition Poor
Keywords: obesity; overweight; food insecurity; food assistance program; minimum wage
MeSH Terms: conditions — Obesity; Malnutrition; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low-Wage Workers from Minneapolis, MN: Low-wage workers from Minneapolis, MN, where the minimum wage will be increased to $15-an-hour over the study period.
  Interventions: Other: Increase Minimum Wage to $15-an-hour
- Low-Wage Workers from Raleigh, NC: Low-wage workers from Raleigh, NC, where the minimum wage will not be significantly changed over the study period.
  Interventions: Other: No Increase in Minimum Wage

INTERVENTIONS:
Other: Increase Minimum Wage to $15-an-hour — Increase in minimum wage to $15-an-hour
  Groups: Low-Wage Workers from Minneapolis, MN
Other: No Increase in Minimum Wage — No increase in minimum wage
  Groups: Low-Wage Workers from Raleigh, NC

SUMMARY:
To evaluate the effect of the Minneapolis minimum wage ordinance on change in body mass index among low-wage workers.

DETAILED DESCRIPTION:
On June 30 2017, Minneapolis became the 40th local jurisdiction to set the minimum wage above the state level, following a succession of other cities and counties across the U.S that have passed similar ordinances since 2012. The city of Minneapolis will incrementally increase the minimum wage from $9.50 to $15 by July 1, 2022 for all businesses with greater than 100 employees; minimum wage in smaller businesses will increase from $7.75 to $13.50 during this same time period. The ordinance specifically states that its purpose is to "maintain worker's health, efficacy, and general well-being." A report by members of the study team at the Humphrey School of Public Affairs at University of Minnesota estimates that the ordinance would increase wages by an average of 22% for the 71,000 city workers making minimum wage or just above minimum wage; moreover, it would affect 41% of non-Hispanic black workers and 54% of Hispanic workers, compared with 17% of white workers. The report also projects a post-policy decrease in food insecurity of 3.8 percentage points and an increase in food expenditures of $26 per week among affected workers.

The available evidence suggests that minimum wage laws may be associated with a range of health outcomes, including obesity. Obesity affects 36.5% of Americans, and is disproportionately high among non-Hispanic blacks and Hispanics. A study by Meltzer and Chen (2009) estimated that 10% of the increase in body mass in the U.S. since 1970 can be explained through the diminished value of minimum wages by inflation, while Kim & Leigh (2010) used instrumental variables to demonstrate that low wages increase the risk of obesity. Mechanisms through which increasing the minimum wage could reduce obesity include improving food security and reducing cost constraints for purchasing healthier foods. However, existing studies linking wages and weight have design weaknesses that limit causal inference and the ability to identify causal mechanisms. A prospective study with a strong counterfactual condition is needed to test whether and how an increase in minimum wage results in improved obesity-related outcomes among low-wage workers.

Throughout the 4.5-year implementation period of the Minneapolis minimum wage ordinance (January 1, 2018-July 1, 2022), the team will follow a cohort of low-wage workers in a natural experiment, using a difference-in-difference design to compare a panel of obesity-related measures among low-wage workers (those earning ≤$10 an hour at baseline) in Minneapolis (n = 400) with low-wage workers in a comparison city with no minimum wage increase (Raleigh, North Carolina, n = 400).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Plan to serve in the workforce for at least 5 years
* Have an address and phone number where they can receive mail and phone calls (though they do not necessarily need to own a phone or have a permanent home)
* Speak English or Spanish well enough to complete the survey
* Either A OR B must be true:

A: Work at a wage of $11.50 an hour for at least an average of 10 hours a week, with at least 2 of those hours at a job in Minneapolis B: Be currently unemployed, but worked at a wage of $11.50 an hour or less for at least an average of 10 hours a week in the last 6 months AND be currently looking for working in Minneapolis

Exclusion Criteria:

* Federal or state workers
* Full-time students
* Plan to retire or move more than 100 miles away in the next 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low wage workers living in Minneapolis, MN or Raleigh, NC.
Sampling Method: Non-Probability Sample
Enrollment: 974 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index | 5 years
  Body mass index (BMI) will be measured over 5 years among low-wage workers in Minneapolis compared to workers in a comparison (control) city, as assessed by objective annual height and weight measurements.

SECONDARY OUTCOMES:
Change Purchase of Healthier Foods | 5 years
  Change in purchasing of healthier foods (e.g. fruits and vegetables) and less healthy foods (e.g. sugar sweetened beverages) will be measured by 2 weeks of food purchase receipts, among a cohort of low-wage workers in Minneapolis compared to a control city.
Change in Food Insecurity | 5 years
  Change in food insecurity will be measured by the U.S. Household Food Security Survey Module: Six-Item Short Form (from the Economic Research Service, USDA September 2012), among a cohort of low-wage workers in Minneapolis compared to a control city. Scores are calculated by simple addition for the 6 items. Scores range from 0 (high food security) to 6 (very low food security).
Change in Food Assistance Program Participation | 5 years
  Change in participation in government-supported food assistance program (SNAP, WIC, FRPL) will be measured by self report among a cohort of low-wage workers in Minneapolis compared to a control city.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin E Caspi, ScD, Principal Investigator — University of Connecticut
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No